CLINICAL TRIAL: NCT00846040
Title: Selective Reduction of Dietary Carbohydrate Versus Fat: Effects on Metabolism, Endocrine Physiology, Brain Activity and Reward Circuitry
Brief Title: Reduced Carbohydrate Versus Fat in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 090081; 09-DK-0081 (Other: NIDDK/NIH)
Record Dates: First submitted 2009-02-14; First posted 2009-02-18 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-01-22

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Carbohydrate; Fat; Macronutrient Balance; Healthy Volunteer
MeSH Terms: conditions — Obesity; Weight Loss; Platelet Glycoprotein IV Deficiency | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Obese RF then RC (Experimental): Obese adult volunteers (BMI above 30 kg/m2) randomized to receive an 85% reduction of baseline dietary fat (RF) for 2 weeks. After a washout period of 2 weeks, they then received a 60% reduction of baseline dietary carbohydrate (RC) for 2 weeks
  Interventions: Other: Reduced fat diet; Other: Reduced carbohydrate diet; Drug: Drug: f-18 fallypride; Device: fMRI; Device: PET
- Obese RC then RF (Experimental): Obese adult volunteers (BMI above 30 kg/m2) randomized to receive a 60% reduction of baseline dietary carbohydrate (RC) for 2 weeks. After a washout period of 2 weeks, they then received an 85% reduction of baseline dietary fat (RF) for 2 weeks.
  Interventions: Other: Reduced fat diet; Other: Reduced carbohydrate diet; Drug: Drug: f-18 fallypride; Device: fMRI; Device: PET
- Lean Control (Active Comparator): Lean adult volunteers (BMI below 30kg/m2) placed on a weight-maintenance diet using a standard diet composition of 50% carbohydrate, 35% fat, and 15% protein on an out-patient basis
  Interventions: Drug: Drug: f-18 fallypride; Device: fMRI; Device: PET

INTERVENTIONS:
Other: Reduced fat diet — RF (selective reduction of 85% of baseline fat calories per day)
  Arms: Obese RC then RF; Obese RF then RC
Other: Reduced carbohydrate diet — RC (selective reduction of 60% of baseline carbohydrate calories per day)
  Arms: Obese RC then RF; Obese RF then RC
Drug: Drug: f-18 fallypride — Dopamine D2 receptor availability is measured by positron emission tomography (PET) using the positron emitting compound [18F] fallypride which binds competitively with dopamine to the D2 receptor.
Device: fMRI — Functional MRI (fMRI) will be used to measure the effects of diet and weight loss on regional brain activity
  Other Names: Functional MRI
Device: PET — Positron emission tomography (PET) will be used to assess whether To assess whether brain activity and reward pathways are altered
  Other Names: Positron emission tomography

SUMMARY:
Popular weight loss strategies often involve reducing an individual's consumption of carbohydrates or fat. However, no controlled study has been carried out to evaluate the effects of reducing carbohydrate versus fat consumption while keeping the other nutrients at standard levels to maintain an individual's weight. Researchers are interested in investigating how different restrictions of carbohydrates or fats affect the many processes involved in weight loss, including brain activity and blood and brain chemical composition.

DETAILED DESCRIPTION:
Popular weight loss strategies often prescribe a targeted reduction of dietary carbohydrate or fat. But surprisingly, no controlled human feeding study has ever investigated the effects of a selective reduction of dietary carbohydrate versus fat while keeping the other dietary macronutrients at their baseline weight-maintenance values. The present study was designed to address this knowledge gap and improve our understanding of how selective reduction of dietary fat versus carbohydrate may differentially impact the many feedback control processes that act to resist weight loss.

Objectives:

- To determine the comparative effects of two controlled fat- or carbohydrate-restricted diets and an outpatient weight loss program on blood and brain chemical composition, weight loss (fat and lean body mass), and regional brain activity in lean and obese individuals.

Eligibility:

- Healthy individuals between 18 and 45 years of age who are either lean (body mass index between 18.5 kg/m(2) and 25 kg/m(2)) or obese (body mass index above 30.0 kg/m(2), weight less than 350 pounds) and are right-handed.

Design:

* Lean participants: Participants will be screened with a medical history, physical examination, blood and urine tests, and weight maintenance observations (food diaries and physical activity monitors). For the scanning visit, participants will receive balanced meals from the National Institutes of Health to consume for 2 days before the visit. During the scanning visit, participants will continue to eat the weight maintenance diet, complete questionnaires, and have a series of imaging studies (including positron emission tomography and magnetic resonance imaging tests) to evaluate brain response to food and other stimuli.
* Obese participants: Participants will be screened with a medical history, physical examination, blood and urine tests, and weight maintenance observations (food diaries and physical activity monitors). During the first inpatient visit, obese participants will eat a weight-maintenance diet for 5 days to establish baseline measurements. After several days of eating a weight-maintenance diet, 20 obese adult volunteers (BMI above 30 kg/m2) will be admitted to the metabolic clinical research unit (MCRU) and, after 5 additional days of the baseline diet, their diets will be modified to result in either 85% reduction of the baseline dietary fat or a 60% reduction of the baseline dietary carbohydrate for the next 6 days. These diet modifications produce an equivalent caloric reduction. The primary outcome measurements will be changes of metabolism, brain reward circuitry and regional brain activity in response to food stimuli measured during the baseline and reduced calorie diet phases. Immediately following each controlled diet, we will measure 3 days of ad-libitum food intake using a computerized vending machine system. The subjects will return to the MCRU after a 2-10 week washout period to receive the opposite reduced calorie diet. Twenty control subjects with normal body weight (BMI between 18.5 - 25 kg/m2) will have measurements of brain reward circuitry and regional brain activity in response to food stimuli while on a balanced, weight-maintenance diet. Immediately following the second in-patient visit, all of the obese subjects will be assigned to a 12 week out-patient weight loss program with the goal of achieving at least 5% weight loss. We will investigate the relationship between short-term fat imbalances measured during the in-patient phases, and the body weight and fat changes during the weight loss program. We will evaluate the effects of weight loss on metabolism, brain reward circuitry, and regional brain activity in response to food stimuli. Finally, if the subjects are available for long-term follow-up, then we will investigate their metabolic phenotype, brain reward circuitry, and regional brain activity in response to food stimuli yearly over the subsequent 5 years following the weight loss intervention. This study will result in an improved understanding of the physiological mechanisms that sense and respond to negative energy balance acutely, after several weeks, and after several years, and may eventually lead to increased long-term success of obesity treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-45 years, male or female
* Body mass less than 350 lbs. (max. weight dictated by table limit for functional magnetic resonance imaging (fMRI) scanner) when acquisition of large bore fMRI is complete, max. wt. limit will increase to 400 lbs.
* Weight stable (less than plus or minus 5 kg over past 6 months)
* Body mass index greater than or equal to 30.0 kg/m(2)
* Premenopausal (women only)
* Healthy, as determined by medical history and laboratory tests
* Able to complete daily bouts of walking at a moderate rate
* Written informed consent

EXCLUSION CRITERIA:

* Body mass greater than 350 lbs. (max. weight dictated by table limit for fMRI scanner) when acquisition of large bore fMRI is complete, max. wt. limit will increase to 400 lbs.
* BMI less than 30.0 kg/m(2)
* Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, diabetes, thyroid disease)
* Taking any prescription medication (except birth control) or other drug that may influence metabolism (e.g. diet/weight-loss medication)
* Hematocrit less than 34% (women only)
* Hematocrit less than 40% (men only)
* Pregnancy, lactation (women only)
* Allergy to lidocaine or ethanol
* Participating in a regular exercise program (greater than 2h/week of vigorous activity)
* Caffeine consumption greater than 150 mg/day (will be clamped at baseline intake during study)
* Regular use of alcohol (greater than 2 drinks per day), tobacco (smoking or chewing), amphetamines, cocaine, heroin, or marijuana over past 6 months
* Past or present history of eating disorder (including binge eating) or psychiatric disease
* Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, multiple food allergies)
* Are claustrophobic to a degree that they would feel uncomfortable in the MRI machine.
* Having any metal in their body (for example, pacemakers, metallic prostheses such as cochlear implants or heart valves, shrapnel fragments, etc.).
* Left-handedness
* Non-native English speakers
* Volunteers unwilling or unable to give informed consent

Control Subjects

INCLUSION CRITERIA:

* Age 18-45 years, male or female
* 18.5 kg/m(2) less than BMI less than 25.0 kg/m(2)
* Weight stable (less than plus or minus 5 kg over past 6 months)
* Premenopausal (women only)
* Healthy, as determined by medical history and laboratory tests
* Written informed consent

EXCLUSION CRITERIA:

* BMI less than 18.5 or greater than 25.0 kg/m(2)
* Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer or diabetes)
* Taking any prescription medication (except birth control) or other drug that may influence metabolism (e.g. diet/weight-loss medication)
* Hyperlipidemia (fasting plasma triglyceride concentration greater than 150 mg/dl)
* Hematocrit less than 34% (women only)
* Hematocrit less than 40% (men only)
* Pregnancy, lactation (women only)
* Participating in a regular exercise program (greater than 2h/week of vigorous activity)
* Caffeine consumption greater than 150 mg/day
* Regular use of alcohol (greater than 2 drinks per day), tobacco (smoking or chewing), amphetamines, cocaine, heroin, or marijuana over the past 6 months
* Past or present history of eating disorder (including binge eating) or psychiatric disease
* Volunteers with strict dietary concerns (e.g vegetarian or kosher diet, multiple food allergies)
* Are claustrophobic to a degree that they would feel uncomfortable in the MRI machine.
* Having any metal in their body (for example, pacemakers, metallic prostheses such as cochlear implants or heart valves, shrapnel fragments, etc.).
* Left-handedness
* Non-native English speakers
* Volunteers unwilling or unable to give informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02-13; Primary Completion 2014-02-24 (Actual); Study Completion 2014-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Allison DB, Zannolli R, Narayan KM. The direct health care costs of obesity in the United States. Am J Public Health. 1999 Aug;89(8):1194-9. doi: 10.2105/ajph.89.8.1194. PMID 10432905
- [Background] Samaha FF, Iqbal N, Seshadri P, Chicano KL, Daily DA, McGrory J, Williams T, Williams M, Gracely EJ, Stern L. A low-carbohydrate as compared with a low-fat diet in severe obesity. N Engl J Med. 2003 May 22;348(21):2074-81. doi: 10.1056/NEJMoa022637. PMID 12761364
- [Result] Hall KD, Bemis T, Brychta R, Chen KY, Courville A, Crayner EJ, Goodwin S, Guo J, Howard L, Knuth ND, Miller BV 3rd, Prado CM, Siervo M, Skarulis MC, Walter M, Walter PJ, Yannai L. Calorie for Calorie, Dietary Fat Restriction Results in More Body Fat Loss than Carbohydrate Restriction in People with Obesity. Cell Metab. 2015 Sep 1;22(3):427-36. doi: 10.1016/j.cmet.2015.07.021. Epub 2015 Aug 13. PMID 26278052
- [Result] Guo J, Simmons WK, Herscovitch P, Martin A, Hall KD. Striatal dopamine D2-like receptor correlation patterns with human obesity and opportunistic eating behavior. Mol Psychiatry. 2014 Oct;19(10):1078-84. doi: 10.1038/mp.2014.102. Epub 2014 Sep 9. PMID 25199919
- [Result] Simmons WK, Rapuano KM, Ingeholm JE, Avery J, Kallman S, Hall KD, Martin A. The ventral pallidum and orbitofrontal cortex support food pleasantness inferences. Brain Struct Funct. 2014 Mar;219(2):473-83. doi: 10.1007/s00429-013-0511-0. Epub 2013 Feb 9. PMID 23397317
- [Result] Simmons WK, Rapuano KM, Kallman SJ, Ingeholm JE, Miller B, Gotts SJ, Avery JA, Hall KD, Martin A. Category-specific integration of homeostatic signals in caudal but not rostral human insula. Nat Neurosci. 2013 Nov;16(11):1551-2. doi: 10.1038/nn.3535. Epub 2013 Sep 29. PMID 24077565
- [Derived] Darcey VL, Guo J, Courville AB, Gallagher I, Avery JA, Simmons WK, Ingeholm JE, Herscovitch P, Martin A, Hall KD. Dietary fat restriction affects brain reward regions in a randomized crossover trial. JCI Insight. 2023 Jun 22;8(12):e169759. doi: 10.1172/jci.insight.169759. PMID 37345661
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-DK-0081.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 71 participants were screened and 43 were enrolled.
Groups:
- Obese RF Then RC: Obese adult volunteers (BMI above 30 kg/m2) randomized to receive an 85% reduction of baseline dietary fat for 2 weeks, then a 60% reduction of baseline dietary carbohydrate for 2 weeks. Each admission starts with a 5 day baseline period before the randomized diet.
- Obese RC Then RF: Obese adult volunteers (BMI above 30 kg/m2) randomized to receive a 60% reduction of baseline dietary carbohydrate for 2 weeks, then an 85% reduction of baseline dietary fat for 2 weeks. Each admission starts with a 5 day baseline period before the randomized diet.
- Lean Control: Lean adult volunteers (BMI below 30kg/m2) placed on a weight-maintenance diet using a standard diet composition of 50% carbohydrate, 35% fat, and 15% protein for 2 days on an out-patient basis followed by an admission to the metabolic unit for 3 days.
Period: Baseline: Days 1-5
Arm/Group | Obese RF Then RC | Obese RC Then RF | Lean Control
Started | 10 | 10 | 23
Completed | 9 | 10 | 23
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: First Treatment Period: Days 6-14
Arm/Group | Obese RF Then RC | Obese RC Then RF | Lean Control
Started | 9 | 10 | 0 (This group participated in only the baseline period)
Completed | 9 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Washout: 2 Weeks to 10 Weeks
Arm/Group | Obese RF Then RC | Obese RC Then RF | Lean Control
Started | 9 | 10 | 0
Completed | 9 | 8 | 0
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Second Treatment: After Washout, 14 Day
Arm/Group | Obese RF Then RC | Obese RC Then RF | Lean Control
Started | 9 | 8 | 0
Completed | 9 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Obese RF Then RC: Obese adult volunteers (BMI above 30 kg/m2) randomized to receive an 85% reduction of baseline dietary fat for 2 weeks, then a 60% reduction of baseline dietary carbohydrate for 2 weeks
- Obese RC Then RF: Obese adult volunteers (BMI above 30 kg/m2) randomized to receive a 60% reduction of baseline dietary carbohydrate for 2 weeks, then an 85% reduction of baseline dietary fat for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Obese RF Then RC | Obese RC Then RF | Lean Control | Total
Number analyzed (Participants) | 10 | 10 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (6.9) | 35.6 (8.1) | 28 (6.2) | 31.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 11 | 21
  Male | 4 | 6 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 23 | 41
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 12 | 26
  White | 3 | 1 | 9 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Quotient (RQ)
Description: Respiratory quotient was calculated as the ratio of carbon dioxide production to oxygen consumption as measured in a metabolic chamber for at least 23 continuous hours on days 2 and 5 of the baseline diet and days 1, 4, and 6 of the reduced-energy diets.
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: ratio
Groups:
- RC Diet: Reduced carbohydrate diet
- RF Diet: Reduced fat diet
Arm/Group | RC Diet | RF Diet
Number analyzed (Participants) | 19 | 17
ratio | -0.0552 (0.003) | 0.00453 (0.003)

2. Secondary Outcome: Change in 24 Hour Energy Expenditure
Description: 24 hour energy expenditure was measured in a respiratory chamber.
Time Frame: Baseline and 14 days
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | RC Diet | RF Diet
Number analyzed (Participants) | 19 | 17
kcal/day | -97.7 (23) | -49.6 (24)

3. Secondary Outcome: Change in Cumulative Fat Imbalance
Description: Measured as the difference between dietary fat intake and fat oxidation by the body as measured in the respiratory chamber
Time Frame: Baseline and 14 days
Measure: Mean (Standard Error); unit: grams
Arm/Group | RC Diet | RF Diet
Number analyzed (Participants) | 19 | 17
grams | -245 (21) | -463 (37)

4. Secondary Outcome: Caudate Dopamine D2-like Receptor Binding Potential (D2BP)
Description: The time-activity curves for [18F]fallypride tracer concentration in the ROIs were measured by PET and kinetic parameters were fit to a four compartment mathematical model (with the cerebellum used as the reference tissue). D2BP was expressed as the dimensionless ratio of rate constants quantifying binding and unbinding of tracer in the regions of interest.
Time Frame: Day 2 of in-patient admission
Measure: Mean (95% Confidence Interval); unit: ratio
Groups:
- Obese: Obese adult volunteers (BMI above 30 kg/m2)
- Lean Control: Lean adult volunteers (BMI below 30kg/m2)
Arm/Group | Obese | Lean Control
Number analyzed (Participants) | 20 | 23
ratio | 28.2 [26.48 to 29.86] | 24.9 [22.95 to 26.92]

5. Secondary Outcome: Putamen Dopamine D2-like Receptor Binding Potential (D2BP)
Description: as for outcome 4
Time Frame: Day 2 of in-patient admission
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Obese | Lean Control
Number analyzed (Participants) | 20 | 23
ratio | 30.7 [28.61 to 32.7] | 27 [25.14 to 28.93]

6. Secondary Outcome: Accumbens Dopamine D2-like Receptor Binding Potential (D2BP)
Description: as for outcome 4
Time Frame: Day 2 of in-patient admission
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Obese | Lean Control
Number analyzed (Participants) | 20 | 23
ratio | 18.3 [16.6 to 19.94] | 16.7 [14.16 to 19.29]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks after the second in-patient visit
Groups:
- Obese Reduced Carbohydrate: Reduced carbohydrate diet (selective reduction of 60% of baseline carbohydrate calories per day)
- Obese Reduced Fat: Reduced fat diet (selective reduction of 85% of baseline fat calories per day)
Arm/Group | Obese Reduced Carbohydrate | Obese Reduced Fat | Lean Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT00846040/Prot_SAP_000.pdf